CLINICAL TRIAL: NCT06295562
Title: Pharmacological Treatment Targeting Endotypic Traits of Obstructive Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Wan-Ju Cheng, Principal Investigator, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH112-REC3-201
Record Dates: First submitted 2024-02-16; First posted 2024-03-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: compensation; upper airway; Taiwan; serotonin; noradrenaline
MeSH Terms: interventions — Atomoxetine Hydrochloride; oxybutynin; Venlafaxine Hydrochloride; Trazodone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- atomoxetine 80mg combined with oxybutynin 5mg (Experimental): Participants will receive atomoxetine 80mg combined with oxybutynin 5mg once (1 h before polysomnographic study).
  Interventions: Drug: Atomoxetine 80mg combined with oxybutynin 5mg; Drug: Placebo
- venlafaxine 37.5mg (Experimental): Participants will receive venlafaxine 37.5mg once (1 h before polysomnographic study).
  Interventions: Drug: Venlafaxine 37.5mg; Drug: Placebo
- atomoxetine 80mg combined with trazodone 100mg (Experimental): Participants will receive atomoxetine 80mg combined with trazodone 100mg once (1 h before polysomnographic study).
  Interventions: Drug: Atomoxetine 80mg combined with trazodone 100mg; Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine 80mg combined with oxybutynin 5mg — Atomoxetine 80mg combined with oxybutynin 5mg
  Arms: atomoxetine 80mg combined with oxybutynin 5mg
Drug: Venlafaxine 37.5mg — Venlafaxine 37.5mg
  Arms: venlafaxine 37.5mg
Drug: Atomoxetine 80mg combined with trazodone 100mg — Atomoxetine 80mg combined with trazodone 100mg
  Arms: atomoxetine 80mg combined with trazodone 100mg
Drug: Placebo — Placebo tablet

SUMMARY:
This study will conduct 3 intervention trials with 44 different participants in each trial, with 22 participants will undergo in-laboratory overnight polysomnograms (PSGs) at one night of medication intervention, and the other 22 at taking placebo (contained starch) 1 h before sleep. Three medication regimens will be tested: (1) atomoxetine 80mg combined with oxybutynin 5mg; (2) venlafaxine 37.5mg; and (3) atomoxetine 80mg combined with trazodone 100mg. Endotypic traits will be estimated using the Phenotyping Using Polysomnography method. The primary outcome is the change in apnea-hypopnea index, and secondary outcomes include endotypic traits and sleep parameters.

ELIGIBILITY:
Inclusion Criteria:

* apnea-hypopnea index ≥ 15 hr-¹

Exclusion Criteria:

* the presence of pulmonary, cardiac, neurologic, or other active severe medical or psychiatric diseases
* current use of continuous positive airway pressure therapy
* use of drugs that might interact with the investigational medication or known to affect sleep during the trial or 1 month before the study
* known allergy to the investigational medication
* current smoking
* heavy alcohol drinking (male > 14 drinks and women >7 drinks per week)
* pregnant or lactating
* periodic limb movement index ≤ 15hr-1
* the presence of sleep-related hypoventilation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Physiological parameter | Baseline and one week
  Change in apnea-hypopnea index.

SECONDARY OUTCOMES:
Endotypic traits | Baseline and one week
  Four endotypic traits, namely arousal threshold, upper airway collapsibility, loop gain, and upper airway muscle compensation, will be estimated using the Phenotyping Using Polysomnography method, specifically, a validated cloud-based Python application (PUPpy).

OTHER OUTCOMES:
Sleep quality | Baseline and one week
  Sleep quality is assessed using a 3-point Likert scale ranging from 1 (very good) to 3 (very poor)
Waking sleepiness | Baseline and one week
  Waking sleepiness is assessed using a 4-point Likert scale ranging from 1 (very sleepy) to 4 (not at all sleepy).

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No